CLINICAL TRIAL: NCT04505007
Title: Guideline-Directed Medical Therapy in Patients After Implantation of Implantable Cardioverter Defibrillators to Improve Long-Term Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ratika Parkash (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Ratika Parkash, Cardiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ICD-GDMT
Record Dates: First submitted 2020-07-23; First posted 2020-08-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: randomized 1:1 to either arm
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Patients will be coded with a unique identifier.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual clinical care (No Intervention): In this arm, patients with devices and heart failure will undergo usual clinical care. This consists of follow-up as deemed necessary by their primary care providers.
- Specialized clinic (Experimental): In this arm, patients with devices and heart failure will be enrolled in a specialized clinic with the following aims:
  1. Referral to a heart failure nurse practitioner to undergo optimization of medical therapy.
  2. Optimization of device programming with reduction of ventricular pacing where possible, rate responsiveness when indicated.
  3. For those patients with CRT - ECG optimization using a previously tested protocol will be performed. This will consist of attempts to achieve the shortest QRS duration with the following guidelines:
     1. Two BV fusion patterns in leads V1 and V2: QRS normalization or a new or an increased R wave.
     2. QRS difference ≤-25 ms. Remodelling probability increases as QRS difference takes on larger negative values (QRS difference = BV paced QRS - LBBB QRS duration, in ms).
  Interventions: Other: Specialized heart function clinic

INTERVENTIONS:
Other: Specialized heart function clinic — This information has already been provided.
  Arms: Specialized clinic

SUMMARY:
Guideline-directed medical therapy (GDMT) and the mortality benefit it provides in the heart failure with reduced ejection fraction (HFrEF) population are well-established by multiple professional society guidelines. GDMT refers to initial medical therapy with angiotensin-converting enzyme inhibitors (ACEi) or angiotensin-receptor blockers (ARB), beta-blockers (BB), and mineralocorticoid receptor antagonists (MRA) titrating to maximally tolerated doses for patients with HFrEF. Cardiac implantable electronic devices (CIEDs) such as the implantable cardioverter defibrillator (ICD) and cardiac resynchronization therapy (CRT) have also become a mainstay in the management of HFrEF after implementation of GDMT. ICD therapy is an effective and established treatment for HFrEF patients for both primary and secondary prevention of SCD.

Regarding the use, adherence and results of GDMT after ICD/CRT implantation, there is very limited data available in the literature. There are a few retrospective trials that show this, however very limited randomized controlled data.

This proposed study would randomize patients with primary prevention ICDs and CRT into a specialized clinic with a heart failure nurse practitioner vs usual clinical care, with the goal of determining outcomes such as change in LVEFs, heart failure hospitalizations, and visits to the ER for heart failure. Consequently, this would determine whether targeted clinics are needed for ICD/CRT patients with HFrEF to optimize GDMT, improve patient outcomes and thus implement new guidelines/recommendations for this specific patient population.

DETAILED DESCRIPTION:
Guideline-directed medical therapy (GDMT) and the mortality benefit it provides in the heart failure with reduced ejection fraction (HFrEF) population are well-established by multiple professional society guidelines. GDMT refers to initial medical therapy with angiotensin-converting enzyme inhibitors (ACEi) or angiotensin-receptor blockers (ARB), beta-blockers (BB), and mineralocorticoid receptor antagonists (MRA) titrating to maximally tolerated doses for patients with HFrEF. Cardiac implantable electronic devices (CIEDs) such as the implantable cardioverter defibrillator (ICD) and cardiac resynchronization therapy (CRT) have also become a mainstay in the management of HFrEF after implementation of GDMT. ICD therapy is an effective and established treatment for HFrEF patients for both primary and secondary prevention of SCD. Canadian guidelines recommend ICD implantation for patients with ischemic or non-ischemic cardiomyopathy (NICM) and persistent ejection fraction ≤ 30%, when persistent refers to at least 3 months of optimal medical therapy (OMT) in all patients and, in patients with ischemic heart disease, at least 3 months after revascularization and at least 40 days after a myocardial infarction (MI). These guidelines also suggest that ICDs be considered for the same population with a left ventricular ejection fraction (LVEF) of 31-35% as well. CRT device therapy is indicated for use in patients in sinus rhythm with New York Heart Association (NYHA) class II-III, or ambulatory NYHA class IV heart failure symptoms, a LVEF ≤ 35%, and QRS duration > 130 ms because of left bundle branch block (LBBB).

The use and adherence to GDMT before and after ICD implantation is of critical importance. Adherence to GDMT before implantation has the potential to improve survival and may even improve left ventricular ejection fraction (LVEF) enough so that an ICD may no longer be indicated. However, adherence to GDMT is notoriously difficult to assess in conventional clinical practice due a multitude of factors. These include information about outpatient prescription use, prescription filling pattern/barriers, reported patient adherence to GDMT, and various electronic health records/documentation linked to pharmacies to name a few. In one retrospective study, it was demonstrated that just over half (61.1%) of patients filled any GDMT prescription before ICD implantation. Futhermore, patients receiving GDMT versus those who did not receive GMT had a lower 1 year mortality rate after ICD implantation (11.1% vs 16.2%) after adjustments for comorbidities, LVEF, and NYHA class heart failure. In a similar study assessing prescriptions claim data to assess beta-blocker use prior to ICD implantation, the median number of days covered by a beta-blocker in the 90 days prior to ICD implantation was 46 days. From the results of these studies, it is clear that there is room for improvement for implementation of GDMT prior to ICD implantation.

Regarding the use, adherence and results of GDMT after ICD/CRT implantation, there is very limited data available in the literature. One of the first studies to exhibit the effect of medical therapy in HFrEF patients after ICD/CRT implantation was a retrospective cohort study that stratified ICD/CRT patients according to combination treatment with HFrEF medical therapy; patients on none or one HFrEF medications were in group 0/1, patients on two HFrEF medications (ex: ACEi + BB) were in group 2, and patients on all three HFrEF medications (ACEi/ARB + BB + MRA) were in group 3. Results showed a higher hospitalization rate per patient/year in the undertreated population (group 0 and 1) (28% vs 12%, p = 0.001). Also, in multivariate analysis, patients treated with better medical therapy (groups 2 and 3) had less hospitalizations for heart failure and better survival (p < 0.001). In addition to benefits with hospitalizations and better survival, adjunctive optimization of GDMT can result in quantitative benefits as well. One study compared usual post-implant care was compared to protocol-driven clinical care with a dedicated nurse and cardiologist. Protocol-driven care was associated with significant improvements in LVEF, LV internal diastolic diameter, and improvements in maximum exercise capacity. Interestingly, these improvements appeared to be driven not only by device-related management, but also by concomitant optimization of GDMT and heart failure education. As evidenced by these promising results, it is of utmost importance to assess and optimize the use of GDMT in patients with CIEDs and HFrEF, as there can be potential improvements in LVEF, exercise capacity and survival.

This proposed study would randomize patients with primary prevention ICDs and CRT into a specialized clinic with a heart failure nurse practitioner vs usual clinical care, with the goal of determining outcomes such as change in LVEFs, heart failure hospitalizations, and visits to the ER for heart failure. Consequently, this would determine whether targeted clinics are needed for ICD/CRT patients with HFrEF to optimize GDMT, improve patient outcomes and thus implement new guidelines/recommendations for this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

- patients who underwent ICD or CRT (pacemaker or defibrillator) implantation therapy at the QEII Health Sciences Centre between 2002 and 2019 and had a left ventricular ejection fraction ≤ 35% at the time of the initial implantation.

Exclusion Criteria:

* unable to provide informed consent, has a life expectancy of less than one year, dementia, cirrhosis, or metastatic malignancy.
* Patients who underwent primary prevention ICD implantation for arrhythmogenic right ventricular cardiomyopathy (ARVC), ion channelopathies, hypertrophic cardiomyopathy, or infiltrative cardiomyopathy will be excluded from this analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | 1 year
  The proportion of patients that experience more than 10% increase in LVEF. This outcome will demonstrate if the experimental group had benefit in their heart function (ie LVEF). A successful outcome is if the patient demonstrated an increase by at least 10% in the LVEF over the year of follow up.

SECONDARY OUTCOMES:
Mortality rate | 1 year
  All-cause mortality will demonstrate if the two groups differed in the absolute number of mortality in the 1 year follow up period.
Heart failure hospitalization frequency | 1 year
  This will determine if the experimental group patients were hospitalized with a different frequency compared to the usual care group during the 1 year follow up period.
Rate of adherence to guideline directed medical therapy | 1 year
  This outcome will be based on self-reported adherence to combinations of medications for treating heart failure. Patients will provide us details of adherence to their medications as best as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD, Principal Investigator — NSHA
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezekowitz JA, O'Meara E, McDonald MA, Abrams H, Chan M, Ducharme A, Giannetti N, Grzeslo A, Hamilton PG, Heckman GA, Howlett JG, Koshman SL, Lepage S, McKelvie RS, Moe GW, Rajda M, Swiggum E, Virani SA, Zieroth S, Al-Hesayen A, Cohen-Solal A, D'Astous M, De S, Estrella-Holder E, Fremes S, Green L, Haddad H, Harkness K, Hernandez AF, Kouz S, LeBlanc MH, Masoudi FA, Ross HJ, Roussin A, Sussex B. 2017 Comprehensive Update of the Canadian Cardiovascular Society Guidelines for the Management of Heart Failure. Can J Cardiol. 2017 Nov;33(11):1342-1433. doi: 10.1016/j.cjca.2017.08.022. Epub 2017 Sep 6. PMID 29111106
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Colvin MM, Drazner MH, Filippatos GS, Fonarow GC, Givertz MM, Hollenberg SM, Lindenfeld J, Masoudi FA, McBride PE, Peterson PN, Stevenson LW, Westlake C. 2017 ACC/AHA/HFSA Focused Update of the 2013 ACCF/AHA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Failure Society of America. Circulation. 2017 Aug 8;136(6):e137-e161. doi: 10.1161/CIR.0000000000000509. Epub 2017 Apr 28. No abstract available. PMID 28455343
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P. [2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure]. Kardiol Pol. 2016;74(10):1037-1147. doi: 10.5603/KP.2016.0141. No abstract available. Polish. PMID 27748494
- [Background] Bennett M, Parkash R, Nery P, Senechal M, Mondesert B, Birnie D, Sterns LD, Rinne C, Exner D, Philippon F, Campbell D, Cox J, Dorian P, Essebag V, Krahn A, Manlucu J, Molin F, Slawnych M, Talajic M. Canadian Cardiovascular Society/Canadian Heart Rhythm Society 2016 Implantable Cardioverter-Defibrillator Guidelines. Can J Cardiol. 2017 Feb;33(2):174-188. doi: 10.1016/j.cjca.2016.09.009. Epub 2016 Oct 6. PMID 28034580
- [Background] Exner DV, Birnie DH, Moe G, Thibault B, Philippon F, Healey JS, Tang AS, Larose E, Parkash R. Canadian Cardiovascular Society guidelines on the use of cardiac resynchronization therapy: evidence and patient selection. Can J Cardiol. 2013 Feb;29(2):182-95. doi: 10.1016/j.cjca.2012.10.006. PMID 23351926
- [Background] Roth GA, Poole JE, Zaha R, Zhou W, Skinner J, Morden NE. Use of Guideline-Directed Medications for Heart Failure Before Cardioverter-Defibrillator Implantation. J Am Coll Cardiol. 2016 Mar 8;67(9):1062-1069. doi: 10.1016/j.jacc.2015.12.046. PMID 26940927
- [Background] Hauptman PJ, Swindle JP, Masoudi FA, Burroughs TE. Underutilization of beta-blockers in patients undergoing implantable cardioverter-defibrillator and cardiac resynchronization procedures. Circ Cardiovasc Qual Outcomes. 2010 Mar;3(2):204-11. doi: 10.1161/CIRCOUTCOMES.109.880450. Epub 2010 Mar 2. PMID 20197509
- [Background] Massoullie G, Chouki C, Mulliez A, Rossignol P, Ploux S, Pereira B, Reuillard A, Jean F, Andronache M, Eschalier A, Motreff P, Clerfond G, Bordachar P, Authier N, Eschalier R. Effect of Optimization of Medical Treatment on Long-Term Survival of Patients With Heart Failure After Implantable Cardioverter Defibrillator and Cardiac Resynchronization Device Implantation (from the French National EGB Database). Am J Cardiol. 2018 Mar 15;121(6):725-730. doi: 10.1016/j.amjcard.2017.12.013. Epub 2018 Jan 3. PMID 29402420
- [Background] Mullens W, Kepa J, De Vusser P, Vercammen J, Rivero-Ayerza M, Wagner P, Dens J, Vrolix M, Vandervoort P, Tang WH. Importance of adjunctive heart failure optimization immediately after implantation to improve long-term outcomes with cardiac resynchronization therapy. Am J Cardiol. 2011 Aug 1;108(3):409-15. doi: 10.1016/j.amjcard.2011.03.060. Epub 2011 May 6. PMID 21550578
- [Background] Januzzi JL, Butler J, Fombu E, Maisel A, McCague K, Pina IL, Prescott MF, Riebman JB, Solomon S. Rationale and methods of the Prospective Study of Biomarkers, Symptom Improvement, and Ventricular Remodeling During Sacubitril/Valsartan Therapy for Heart Failure (PROVE-HF). Am Heart J. 2018 May;199:130-136. doi: 10.1016/j.ahj.2017.12.021. Epub 2018 Feb 13. PMID 29754651